CLINICAL TRIAL: NCT03885388
Title: Women's Hospital, Zhejiang University School of Medicine
Brief Title: Combination of Methotrexate(MTX) and Actinomycin(ACTD) in the Low Risk Gestational Trophoblastic Neoplasma （GTN） Patients With Score of 5-6
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Collaborators: Huazhong University of Science and Technology (Other); Qilu Hospital of Shandong University (Other); West China Second University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSEM 13b
Record Dates: First submitted 2019-03-18; First posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Gestational Trophoblastic Tumor; Effects of Chemotherapy; Drug Toxicity
Keywords: GTN; MTX; ACTD
MeSH Terms: conditions — Gestational Trophoblastic Disease; Drug-Related Side Effects and Adverse Reactions | interventions — Methotrexate

STUDY DESIGN:
Intervention Model Description: treatment by combination of methotrexate and actinomycin
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control arm (Active Comparator): single methotrexate multicourse treatment MTX:MTX 0.4mg/kg•d, intramuscular, every two weeks
  Interventions: Drug: MTX
- experimental arm (Experimental): combination of methotrexate and actinomycin multicourse treatment, every two weeks MTX+ACTD:Act-d 0.6mg/m2 Day1,2 intravenous (IV) MTX 100mg/m2 IV Day1(after Act-d) MTX 200mg/m2 Ivgtt Day1(after MTX,500mlNS)
  Interventions: Drug: MTX+ACTD

INTERVENTIONS:
Drug: MTX — multicourse methotrexate chemotherapy
  Other Names: methotrexate
  Arms: control arm
Drug: MTX+ACTD — combination use of methotrexate and actinomycin
  Other Names: methotrexate+actinomycin
  Arms: experimental arm

SUMMARY:
In this study, a prospective, multicenter randomized controlled study was conducted to compare the clinical efficacy and toxicity response of combination MTX+ACTD multi-course regimen in low-risk GTN patients with score 5-6 with standard MTX single-drug multi-course regimen.

DETAILED DESCRIPTION:
The improved prognostic scoring system has been in use for more than 20 years in GTN patients. However, there are also more and more clinical evidences showing that the International Federation of Obstetrics and Gynecology（FIGO）/world health organization (WHO) system is not so perfect. The main problem is that a considerable number of patients are resistant to initial chemotherapy, 25-35% occur in low risk (≤ 6 points), and 70-80% occur in patients with a score of 5-6 points. According to reference, the drug resistance factors include high HCG level before chemotherapy, metastatic foci, histological diagnosis of choriocarcinoma, etc. However, according to the score before 2000, there is a moderate risk score group with 4-6 points, i.e. most of the single drug resistance to the initial regimen occurs in the previous moderate risk score group.Therefore, most scholars believe that there are grey areas with a score of 5-6. According to the analysis of 5-6 scores in the scoring system, the prognosis of single-drug chemotherapy is poor, and the initial remission rate is only about 30-40%. Therefore, many authors call for the current staging scoring system to be revised to a more accurate model so that some patients who may be drug resistant can adopt more effective plans at the beginning of treatment.

In this study, the investigators plan to conduct a prospective, multicenter randomized controlled study to compare the clinical efficacy and toxicity response of combination MTX+ACTD multi-course regimen in low-risk GTN patients with score 5-6 with standard MTX single-drug multi-course regimen. The experiment arm of the trial is multi-course combination of MTX and ACTD. The primary endpoint is complete remission rate of primary treatment or failure of primary treatment. Drug toxicity is surveillanced.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of gestational trophoblastic tumor;
* Patients with prognosis score of 5 and 6
* Primary chemotherapy (preventive chemotherapy is not included);
* Physical strength grade: Karnofsky score ≥ 60;
* WBC ≥ 3.5× 109/L, ANC ≥ 1.5× 109/L, PT ≥ 80× 109/L, serum bilirubin ≤ 1.5 times of normal high limit, transaminase ≤ 1.5 times of normal high limit, BUN, Cr≤ normal;
* Follow-up and good compliance;
* Sign the informed consent form.

Exclusion Criteria:

* Pathological diagnosis is intermediate trophoblastic tumor, including PSTT and ETT；
* There are serious or uncontrollable medical diseases, which are not suitable for chemotherapy;
* Those who receive clinical trials of other drugs at the same time.
* Those who receive Chinese medicine.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-03-08 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
primary complete remission | 24 weeks
  complete remission rate by primary treatment

CONTACTS AND LOCATIONS:
Overall Officials: Weiguo Lu, MD., Study Chair — Women's Hospital, College of Medicine Zhejiang University
Locations (1):
- Weiguo Lv, Hangzhou, Zhejiang, China